CLINICAL TRIAL: NCT04778540
Title: Online Survey of Nutritional Status and Dietary Intakes in Chinese Non-hospitalized Patients With Cancer
Brief Title: Online Survey of Nutrition Status in Chinese Non-hospitalized Cancer Patients
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yu Kang, MD, Professor, Peking Union Medical College Hospital
Other Study IDs: Online-Nutr-Cancer 2021
Record Dates: First submitted 2021-02-25; First posted 2021-03-03 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Survey; Nutrition Status; Cancer Patient
Keywords: Nutrition status; Cancer; Discharged patients; online survey
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a national-wide online survey, which aims to investigate the nutritional status and dietary intakes in Chinese discharged patients with cancer. It will provide relevant data for the "White Paper on Nutritional Diet of Cancer Patients in China", and also provide reference for the relevant work of nutrition support for cancer patients in clinical practice.

DETAILED DESCRIPTION:
Nutritional status has significant impact on clinical outcome and quality of life in patients with cancer. Current surveys show that about 30-80% of patients with cancer have nutritional risk and/or malnutrition, and about 20% of the patients' death are directly caused by malnutrition. Appropriate and standardized nutrition therapy might not only improve the nutritional status, but also the clinical outcomes of patients with cancer, and improve their life quality and dignity.

At present, there is still lack of large-scale investigation and research on nutritional status and dietary intakes in discharged patients with cancer in China, and thus affects the overall level of nutritional management for cancer patients, as well as the formation of related guideline.

Therefore, we will conduct a national-wide cross-sectional online survey, which aim to investigate relevant data of nutritional status and dietary intakes among discharged patients with cancer. Data will be collected through an online semi-structured questionnaire using WeChat forms with a consent form. The link to the questionnaire was sent through emails, WeChat App groups, and other social media. The participants were encouraged to roll out the survey, and send the link to more patients as they could. On receiving and clicking the link, the participants will be directed to the information about the study and informed consent. After they accept to take the survey, they will fill up the demographic details and answer a set of questions related to nutritional status and dietary intake investigation.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of cancer Must be able to use WeChat or related social media Fully understood and voluntarily signed the informed consent

Exclusion Criteria:

Hospitalized patients Pregnant and lactating women Be known to have any psychiatric illness Refused to share the data or no network condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The populations of the discharged patients with cancer who fulfilled the inclusion criteria and agreed to participate in the online survey will be included in this study.
Sampling Method: Probability Sample
Enrollment: 6685 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
the prevalence of nutritional risk | baseline
  the prevalence of nutritional risk according to NRS-2002 criteria
the prevalence of dietary reduction and weight loss | baseline
  the the prevalence of dietary reduction and weight loss

SECONDARY OUTCOMES:
nutrition support of discharged cancer patients | baseline
  the description of nutrition support methods of Chinese discharged cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Kang Yu, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No